CLINICAL TRIAL: NCT00577031
Title: Open-label, Efficacy and Safety Study of Bevacizumab (Avastin®) in Combination With XELOX (Oxaliplatin Plus Xeloda®) for the First-line Treatment of Patients With Metastatic Cancer of the Colon or Rectum - 'OBELIX'
Brief Title: OBELIX Study: A Study of Avastin (Bevacizumab) in Combination With XELOX in Patients With Metastatic Cancer of the Colon or Rectum.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21380
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Oxaliplatin; Drug: Xeloda

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg iv on day 1 of each 3 week cycle
Drug: Oxaliplatin — 130mg/m2 iv on day 1 of each 3 week cycle
Drug: Xeloda — 1000mg/m2 po bid on days 1-14 of each 3 week cycle

SUMMARY:
This single arm study will evaluate the efficacy and safety of a first-line regimen of Avastin and XELOX (oxaliplatin + Xeloda) in patients with metastatic cancer of the colon or rectum. Patients will receive 21-day cycles of treatment, comprising Avastin 7.5mg/kg iv on day 1, oxaliplatin 130mg/m2 iv on day 1, and Xeloda 1000mg/m2 po twice daily on days 1-14, for a maximum of 6 months. Patients with stable disease or complete or partial response may continue on Avastin therapy. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* locally advanced or metastatic colorectal cancer;
* no previous treatment with chemotherapy for metastatic disease;
* at least one measurable lesion.

Exclusion Criteria:

* radiotherapy to any site within 4 weeks before study;
* untreated brain metastases or primary brain tumors;
* clinically significant cardiovascular disease;
* chronic daily treatment with high dose aspirin (>325 mg/day);
* other co-existing malignancies or malignancies diagnosed within last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- Italy (32):
  - Bologna
  - Brescia
  - Cagliari
  - Caserta
  - Catanzaro
  - Cefalù
  - Fano
  - Florence
  - Frattaminore
  - Grosseto
  - Ivrea
  - Latisana
  - Lecce
  - Legnago
  - Legnano
  - Macerata
  - Napoli
  - Negrar
  - Orbassano
  - Padua
  - Palermo
  - Pavia
  - Reggio Calabria
  - Reggio Emilia
  - Rionero in Vulture
  - Roma
  - Salerno
  - San Giovanni Rotondo
  - Sondrio
  - Taormina
  - Torino
  - Verbania

REFERENCES:
- [Derived] Antonuzzo L, Giommoni E, Pastorelli D, Latiano T, Pavese I, Azzarello D, Aieta M, Pastina I, Di Fabio F, Bertolini A, Corsi DC, Mogavero S, Angelini V, Pazzagli M, Di Costanzo F. Bevacizumab plus XELOX as first-line treatment of metastatic colorectal cancer: The OBELIX study. World J Gastroenterol. 2015 Jun 21;21(23):7281-8. doi: 10.3748/wjg.v21.i23.7281. PMID 26109816

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab: Cycles 1-8 (3-week cycles): Participants received bevacizumab 7.5 milligrams per kilogram (mg/kg) intravenously (IV) and oxaliplatin 130 mg per square meter (mg/m^2) IV on Day 1 and capecitabine 1000 mg/m^2 tablets, orally, every 12 hours starting the evening of Day 1 for 14 days continuously; cycle was repeated until disease progression or for a maximum of 8 cycles.
  Cycle 9 and beyond (3-week cycles): If the first 8 cycles were tolerated with no disease progression, participants received bevacizumab 7.5 mg/kg IV on Day 1; the cycle was repeated until disease progression.
Period: Overall Study
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab
Started | 205
Completed | 0
Not Completed | 205
Not completed — Adverse Event | 52
Not completed — Progression of disease | 93
Not completed — Protocol Violation | 5
Not completed — Participant withdrew consent | 13
Not completed — Participant non-compliance | 5
Not completed — Need for surgery | 17
Not completed — Medical decision | 14
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Population: Safety population: all enrolled participants who received at least 1 dose of all study medications.
Groups:
- Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab: Cycles 1-8 (3-week cycles): Participants received bevacizumab 7.5 mg/kg IV and oxaliplatin 130 mg/m^2 IV on Day 1 and capecitabine 1000 mg/m^2 tablets, orally, every 12 hours starting the evening of Day 1 for 14 days continuously; cycle was repeated until disease progression or for a maximum of 8 cycles.
  Cycle 9 and beyond (3-week cycles): If the first 8 cycles were tolerated with no disease progression participants received bevacizumab 7.5 mg/kg IV on Day 1; the cycle was repeated until disease progression.
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.25 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 111

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS): Percentage of Participants With Progressive Disease or Death
Description: PFS was defined as the time period in months from the start of study treatment to the first observation of disease progression or death from any cause, whichever occurred first. Data for participants with no tumor assessments after baseline but who were still alive at the time of the clinical cutoff were censored at Day 1. Participants who underwent surgery after experiencing a sufficient shrinkage of the tumor, had any relapse, new occurrence of colorectal cancer, or who died were all considered as having had an event. Participants who underwent surgery without any such event were censored at the date of the last tumor assessment that documented neither a relapse nor a new colorectal cancer had occurred. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20 percent (%) increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Baseline and Day 1 of every cycle until disease progression or death up to 5 years
Population: Intent-to-treat (ITT) population: all enrolled participants who received at least 1 dose of all study medications and had at least 1 measurable lesion according to the Response Evaluation Criteria In Solid Tumours (RECIST) criteria.
Measure: Number; unit: percentage of participants
Groups:
- Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab: Cycles 1-8 (3-week cycles): Participants received bevacizumab 7.5 mg/kg IV) and oxaliplatin 130 mg mg/m^2 IV on Day 1 and capecitabine 1000 mg/m^2 tablets, orally, every 12 hours starting the evening of Day 1 for 14 days continuously; cycle was repeated until disease progression or for a maximum of 8 cycles.
  Cycle 9 and beyond (3-week cycles): If the first 8 cycles were tolerated with no disease progression participants received bevacizumab 7.5 mg/kg IV on Day 1; the cycle was repeated until disease progression.
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
percentage of participants | 50.25

2. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) Among Participants in the ITT Population Who Had at Least 1 Post-Baseline Assessment
Description: The percentage of participants with a best overall response of CR or PR according to RECIST. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis less than [<]10 millimeters [mm]). No new lesions. PR was defined as a greater than or equal to (≥) 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 9 weeks (every 3 cycles) until end of treatment, disease progression, or withdrawal up to 5 years
Population: Subset of participants in the ITT population who had at least 1 post-baseline tumor assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 165
percentage of participants | 58.79

3. Secondary Outcome: Percentage of Participants With a CR or PR Among Participants in the ITT Population
Description: CR and PR were defined using RECIST v1.0. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis <10 mm). No new lesions. PR was defined as a ≥30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 9 weeks (every 3 cycles) until end of treatment, disease progression, or withdrawal up to 5 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
percentage of participants | 49.24

4. Primary Outcome: PFS: Time to Event
Description: PFS was defined as the time period in months from the start of study treatment to the first observation of disease progression or death from any cause, whichever occurred first. Data for participants with no tumor assessments after baseline but who were still alive at the time of the clinical cutoff were censored at Day 1. Participants who underwent surgery after experiencing a sufficient shrinkage of the tumor, had any relapse, new occurrence of colorectal cancer, or who died were all considered as having had an event. Participants who underwent surgery without any such event were censored at the date of the last tumor assessment that documented that neither a relapse nor a new colorectal cancer had occurred. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Baseline and Day 1 of every cycle until disease progression or death up to 5 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
months | 9.70 [8.43 to 10.49]

5. Secondary Outcome: Time to CR or PR Overall Response - Time to Event
Description: Time to overall response (CR or PR) was calculated as the time between the date of start of treatment until first documented response (CR or PR defined per RECIST v1.0). Participants who did not achieve CR or PR were censored at the date of progression, death, or at last adequate tumor assessment date. Median time to CR or PR overall response was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks (every 3 cycles) until end of treatment, disease progression, or withdrawal up to 5 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
months | 3.93 [2.56 to 4.66]

6. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR or PR During First Line Treatment
Description: CR and PR were defined using RECIST v1.0 criteria. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis <10 mm). No new lesions. PR was defined as a ≥30% decrease under baseline of the sum of diameters of all target lesions. Short axis was used in sum for target nodes, while longest diameter was used in sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 3 weeks (every cycle) to disease progression or death up to 5 years
Population: ITT population, only those participants who achieved a best overall response of CR or PR during first line treatment were included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab: Cycles 1-8 (3-week cycles): Participants received bevacizumab 7.5 mg/kg IV and oxaliplatin 130 mg/m^2 IV on Day 1 and capecitabine 1000 mg/m^2 tablets, orally, every 12 hours starting the evening of Day 1 for 14 days continuously; cycle was repeated until disease progression or for a maximum of 8 cycles.
  Cycle 9 and beyond (3-week cycles):If the first 8 cycles were tolerated with no disease progression participants received bevacizumab 7.5 mg/kg IV on Day 1; the cycle was repeated until disease progression.
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 97
percentage of participants | 54.64

7. Secondary Outcome: Duration of Overall Response Among Participants Whose Best Response Was CR or PR During First Line Treatment - Time to Event
Description: For participants with a best overall response of CR or PR, the duration of overall response was measured from the time that the criteria for CR or PR (whichever occurred first) was met until the first date that progressive disease was objectively documented or until the date of death due to underlying cancer, whichever occurred first. Data for participants who did not have an event or who were alive without an objectively documented progressive disease were censored at the date of last adequate tumor assessment. Median duration of overall response was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 3 weeks (every cycle) to disease progression or death up to 5 years
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 97
months | 8.52 [7.28 to 10.33]

8. Secondary Outcome: Percentage of Participants With a Stable Response During First Line Treatment
Description: Stable response defined as participants with a best overall response of CR, PR, or stable disease (SD), defined using RECIST v1.0 criteria. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis <10 mm). No new lesions. PR was defined as a ≥30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. SD defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: Baseline, every 3 weeks (every cycle) to disease progression or death up to 5 years
Population: ITT population, only participants who achieved a best overall response of CR, PR, or SD during first line treatment were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 152
percentage of participants | 52.63

9. Secondary Outcome: Duration of Stable Response
Description: For participants with a best overall response of CR, PR, or SD during first line treatment, the duration of stable response was measured from the time that the criteria for CR, PR, or SD (whichever occurred first) was met until the first date that progressive disease was objectively documented or until the date of death due to underlying cancer, whichever occurred first. Data for participants who did not have an event or who were alive without an objectively documented progressive disease were censored at the date of last adequate tumor assessment. Median duration of stable response was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 3 weeks (every cycle) to disease progression or death up to 5 years
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 152
months | 10.39 [9.02 to 11.44]

10. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment-failure was defined as discontinuation of treatment for any reason, including the following qualifying events: death due to any cause, adverse event, insufficient therapeutic response (progression of disease), failure to return (lost to follow-up), refusing treatment (participant non-compliance), being unwilling to cooperate and withdrawing consent (participant withdrew consent).
Time Frame: Baseline, every 3 weeks (every cycle) to disease progression or death up to 5 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
percentage of participants | 82.74

11. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment-failure was defined as the time from the first day of treatment to discontinuation of treatment for any reason, including: death due to any cause, adverse event, insufficient therapeutic response (progression of disease), failure to return (lost to follow-up), refusing treatment (participant non-compliance), being unwilling to cooperate and withdrawing consent (participant withdrew consent). For participants who did not experience a qualifying event, their data were censored at the earlier of either the date of last tumour assessment or the date of the last intake of study medication. Median time to treatment-failure was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 3 weeks (every cycle) to disease progression or death up to 5 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
months | 6.69 [5.97 to 7.74]

12. Secondary Outcome: Overall Survival: Percentage of Participants That Died Due to Any Cause
Description: Overall survival was defined as the time from the date of the first day of treatment until the date of death from any cause. If a participant was not known to have died, survival was censored at the last date the participant was known to be alive.
Time Frame: Baseline, Day 1 of every cycle to end-of-treatment, every 3 months during longer-term follow-up, or to death due to any cause up to 5 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
percentage of participants | 50.76

13. Secondary Outcome: Overall Survival: Time to Event
Description: Overall survival was defined as the time from the date of the first day of treatment until the date of death from any cause. If a participant was not known to have died, survival was censored at the last date the participant was known to be alive. Median overall survival was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 12
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 197
months | 23.15 [20.07 to 27.15]

14. Secondary Outcome: Percentage of Participants Undergoing Surgical Intervention With Residual Disease Status Post-surgery
Description: The percentage of participants who underwent surgery during the study period with an evaluation of their disease status after surgery. The surgery during the study period was described by reason: curative, palliative, biopsy, other, or unknown. Residual disease status after surgery was described as: no residual disease due to radical surgery, presence of residual disease, unknown or not applicable.
Time Frame: At surgery, at least 6 to 8 weeks after last dose of bevacizumab up to 5 years
Population: The 52 participant subpopulation of the ITT population who underwent surgery during the time period of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 52
percentage of participants
  Curative, no residual disease | 55.77
  Curative, residual disease | 13.46
  Curative, unknown | 3.85
  Curative, not applicable | 7.69
  Palliative, no residual disease | 3.85
  Palliative, residual disease | 7.69
  Palliative, unknown | 3.85
  Palliative, not applicable | 1.92
  Biopsy, residual disease | 1.92
  Biopsy, not applicable | 1.92
  Unknown, unknown | 1.92
  Unknown, not applicable | 3.85
  Other, residual disease | 1.92
  Other, not applicable | 3.85

15. Secondary Outcome: Percentage of Participants With Best Overall Response of CR or PR by Kirsten Rat Sarcoma Viral Oncogene Homolog (K-Ras)/V-Raf Murine Sarcoma Viral Oncogene Homolog B (B-Raf) Mutation Status
Description: The percentage of participants with a best overall response of CR or PR according to RECIST. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis <10 mm). No new lesions. PR was defined as ≥30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
  The K-Ras and/or the B-Raf gene mutation status of participants was evaluated by the central laboratory using tumor samples. Wild-type participants did not have a mutation in either gene.
Time Frame: Baseline, every 9 weeks (every 3 cycles) until end of treatment, disease progression, or withdrawal up to 5 years
Population: ITT population; only participants with a known K-Ras and/or B-Raf gene mutation status and at least 1 post-baseline tumor assessment. Number (n) equals (=) number of participants with either wild-type or K-Ras/B-Raf gene mutation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 33
percentage of participants
  Wild-type (n=18) | 88.89
  Gene mutation (n=15) | 66.67

16. Secondary Outcome: European Quality of Life 5 Dimension (EQ-5D) Raw-Index Score
Description: Quality of life (QoL) assessments were used to derive pre-specified QoL scores according to the QoL manual "EQ-5D-3 Level (3L)" user guide for instrument version 4.0. The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The visual analog scale (VAS) component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. The overall health score absolute changes were calculated for each participant as follows: (score at the end of treatment minus score at baseline). EQ-5D health states were converted into EQ-5D-3L raw index value by applying the scoring algorithm based on the European EQ-net VAS set. The raw index was chosen instead of rescaled index, since the questionnaire was used in order to obtain a quality of life assessment. The raw index scores ranged from 0 (worst health state) to 100 (best health state).
Time Frame: Baseline, every 9 weeks (every 3 cycles), at end-of-treatment up to 5 years
Population: ITT population, only participants who had EQ-5D-3L scores for both baseline and last visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab
Number analyzed (Participants) | 114
units on a scale
  Baseline | 80.24 (14.32)
  Last visit | 74.94 (19.08)
  Absolute change from baseline | -5.30 (19.13)
Statistical Analysis 1: Comparison: Bevucizamab+Oxaliplatin+Capecitabine/Bevacizumab; Change from baseline to last visit; Test type: Superiority or Other; p = 0.0076, Signed-rank test

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of first administration of study treatment until 28 days after the last dose of study treatment up to 5 years
Groups:
- Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab: Cycles 1-8 (3-week cycles): Participants received bevacizumab 7.5 mg/kg IV) and oxaliplatin 130 mg mg/m^2 IV on Day 1 and capecitabine 1000 mg/m^2 tablets, orally, every 12 hours starting the evening of Day 1 for 14 days continuously; cycle was repeated until disease progression or for a maximum of 8 cycles.
  Cycle 9 and beyond (3-week cycles): If the first 8 cycles were tolerated with no disease progression, participants received bevacizumab 7.5 mg/kg IV on Day 1; the cycle was repeated until disease progression.
Arm/Group | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 56/197
Other Adverse Events (participants affected / at risk) | 179/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab (N=197)
Diarrhoea (Gastrointestinal disorders) | 4
Intestinal obstruction (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 2
Subileus (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Hypersensitivity (Immune system disorders) | 3
Pneumonia (Infections and infestations) | 3
Cachexia (Metabolism and nutrition disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7
Deep vein thrombosis (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 3
Hypertension (Vascular disorders) | 1
Vertebroplasty (Surgical and medical procedures) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal vein thrombosis (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Renal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Oxaliplatin+Capecitabine/Bevacizumab (N=197)
Anaemia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 26
Abdominal pain (Gastrointestinal disorders) | 29
Abdominal pain upper (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 27
Diarrhoea (Gastrointestinal disorders) | 73
Nausea (Gastrointestinal disorders) | 84
Stomatitis (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 48
Asthenia (General disorders) | 60
Fatigue (General disorders) | 29
Mucosal inflammation (General disorders) | 21
Pyrexia (General disorders) | 40
Anorexia (Metabolism and nutrition disorders) | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Headache (Nervous system disorders) | 10
Neuropathy peripheral (Nervous system disorders) | 38
Neurotoxicity (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 59
Proteinuria (Renal and urinary disorders) | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 18
Hypertension (Vascular disorders) | 45
Atrial fibrillation (Cardiac disorders) | 1
Cardiac ventricular disorder (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Dihydropyrimidine dehydrogenase deficiency (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 8
Conjunctivitis (Eye disorders) | 3
Diplopia (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Scleral haemorrhage (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Anal inflammation (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 2
Dental discomfort (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis haemorrhage (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 3
Gingivitis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 4
Inguinal hernia (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 7
Rectal tenesmus (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 5
Discomfort (General disorders) | 1
Facial pain (General disorders) | 1
Hyperpyrexia (General disorders) | 2
Infusion site extravasation (General disorders) | 1
Infusion site pain (General disorders) | 2
Injection site haematoma (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 2
Performance status decreased (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 6
Hypertransaminasaemia (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 4
Hypersensitivity (Immune system disorders) | 4
Bronchitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 2
Herpes virus infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Labyrinthitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 5
Tooth abscess (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 5
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complications (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood iron decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 4
Blood uric acid increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 4
Weight decreased (Investigations) | 8
Weight increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysaesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 9
Migraine (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5
Presyncope (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Syncope vasovagal (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Mood altered (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 4
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Strangury (Renal and urinary disorders) | 2
Balanitis (Reproductive system and breast disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Orchitis noninfective (Reproductive system and breast disorders) | 1
Testicular disorder (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 3
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 5
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 3
Cyst drainage (Surgical and medical procedures) | 1
Aortic thrombosis (Vascular disorders) | 1
Axillary vein thrombosis (Vascular disorders) | 1
Blood pressure fluctuation (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 5
Hot flush (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 5
Lymphoedema (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 4
Thrombophlebitis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 2
Vena cava thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.